CLINICAL TRIAL: NCT03324672
Title: Kinesio Taping and Manual Therapy Efficacity on Lumbar Pain During Pregnancy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI's choice
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TRIGGER
Record Dates: First submitted 2017-10-25; First posted 2017-10-30 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Manual Therapy
Keywords: lumbar pain; pregnancy;
MeSH Terms: conditions — Low Back Pain | interventions — Precipitating Factors

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRIGGER (Active Comparator)
  Interventions: Procedure: TRIGGER
- TRIGGER+CURETAPE (Experimental)
  Interventions: Procedure: TRIGGER+CURETAPE

INTERVENTIONS:
Procedure: TRIGGER — only TRIGGER point will be included for the manual therapy
  Arms: TRIGGER
Procedure: TRIGGER+CURETAPE — TRIGGER point will be included for the manual therapy with kinesio-taping
  Arms: TRIGGER+CURETAPE

SUMMARY:
Pregnant women often suffer from lumbar pain , specially during the last semester . Usually physiotherapy and manual therapy on TRIGGER point help them .

But there is also another type of support , the Kinesio-Taping using the pose of a strip which aims to mobilize the muscle without any restriction.

The purpose is to reduce the pain with the combo therapy (TRIGGER point plus Kinesi Taping)

ELIGIBILITY:
Inclusion Criteria:

* age > 18
* french speaking
* single pregnancy
* lumbar pain
* EIFEL score>6
* medical insurance

Exclusion Criteria:

* twins pregnancy
* rachial arthrodesis
* Probable Acrylique allergy
* Psoriasis or other cutaneous problems
* circulatory disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — only pregnant women
Enrollment: 1 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
French version of Roland-Morris questionnaire in chronic low back pain patients EIFEL Échelle d'Incapacité Fonctionnelle pour l'Évaluation des Lombalgies questionnaire) score | change from week 30 to week 38
  EIFEL questionnaire is filled by patient between week 30 of pregnancy to week 38, scale range from 0 to 24,

SECONDARY OUTCOMES:
Pain scale | change from week 30 to week 38
  Pain scale is filled by patient between week 30 of pregnancay to week 30, scale range from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: AZRIA Elie, MD, Study Director — GHPSJ
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France